CLINICAL TRIAL: NCT00517881
Title: A Single Arm Open Label Study to Assess the Efficacy, Safety and Tolerability of Once Monthly Administration of Subcutaneous C.E.R.A. for the Maintenance of Haemoglobin Levels in Pre-dialysis Patients With Chronic Renal Anaemia
Brief Title: Efficacy, Safety and Tolerability Study of Subcutaneous C.E.R.A. in Pre-Dialysis Participants With Chronic Renal Anemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to the slow recruitment rate.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20944; 2006-006523-40 (EudraCT Number)
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C.E.R.A. (Experimental)
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta (C.E.R.A.)

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta (C.E.R.A.) — Subcutaneous methoxy polyethylene glycol-epoetin beta (C.E.R.A.) at starting dose of 120, 200, or 360 mcg every 4 weeks for 20 weeks. Further dose adjustments will be performed during the study depending on the participant's blood hemoglobin levels.
  Other Names: Mircera

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of subcutaneous methoxy polyethylene glycol-epoetin beta (C.E.R.A.) for maintenance of hemoglobin levels in pre-dialysis participants with chronic renal anemia. Participants currently receiving maintenance treatment with subcutaneous darbepoetin alfa will receive monthly subcutaneous injections of C.E.R.A. with the starting dose of 120, 200 or 360 micrograms (mcg) derived from the dose of darbepoetin alfa or epoetin alfa in the week preceding study start.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal anemia
* Hemoglobin concentration between 10.5 gram per deciliter (g/dL) and 12.5 g/dL
* Adequate iron status (serum ferritin greater than [>] 100 nanogram per milliliter and Transferrin Saturation >20 percent [%] or hypochromic red cells less than [<] 10%)
* Continuous subcutaneous maintenance darbepoetin alfa therapy with same dosing interval during previous 2 months

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months
* Poorly controlled hypertension requiring hospitalization or interruption of darbepoetin alfa treatment in previous 6 months
* Acute or chronic bleeding
* Active malignant disease (except non-melanoma skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Sweden (13):
  - Danderyd
  - Eksjö
  - Eskilstuna
  - Gävle
  - Gothenburg
  - Huddinge
  - Jönköping
  - Kristianstad
  - Skellefteå
  - Stockholm
  - Umeå
  - Värnamo
  - Västervik

RESULTS

PARTICIPANT FLOW:
Groups:
- C.E.R.A.: Participants received subcutaneous methoxy polyethylene glycol-epoetin beta (C.E.R.A.) at starting dose of 120, 200, or 360 micrograms (mcg) every 4 weeks for 20 weeks. Further dose adjustments were performed during the study depending on the participant's blood hemoglobin levels.
Period: Overall Study
Arm/Group | C.E.R.A.
Started | 29
Completed | 24
Not Completed | 5
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 1
Not completed — Renal transplantation | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who were treated with at least 1 dose of the study drug and a safety follow-up, whether withdrawn prematurely or not.
Groups:
- C.E.R.A.: Participants received subcutaneous C.E.R.A. at starting dose of 120, 200, or 360 mcg every 4 weeks for 20 weeks. Further dose adjustments were performed during the study depending on the participant's blood hemoglobin levels.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Mean Hemoglobin Concentration Within Plus or Minus (+/-) 1 Gram Per Deciliter (g/dL) of Their Reference Hemoglobin and Within the Target Range
Description: Percentage of participants maintaining the mean hemoglobin concentration within +/- 1.0 g/dL of their reference hemoglobin value and within the target range of 10.5 to 12.5 g/dL during the efficacy evaluation period (EEP) was reported. The reference hemoglobin value was defined as the mean of the 5 assessments recorded during the stability verification period (SVP) at Weeks -4, -3, -2, -1 and 0. The mean hemoglobin concentration for each individual participant during the EEP (Week 17 to Week 24) was estimated as a time adjusted average.
Time Frame: Week 17 up to Week 24
Population: The Intention-to-treat (ITT) population included all participants who received at least 1 dose of C.E.R.A. (week 0) and for whom data for at least 1 follow-up variable was available. Data missing at the end of the EEP (that is, the last measured hemoglobin value before Week 24) was handled using the last value carried forward method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
percentage of participants | 51.7 [32.5 to 70.6]

2. Secondary Outcome: Change in Hemoglobin Concentration Between Reference (SVP) and EEP
Description: The reference hemoglobin value was defined as the mean of the 5 assessments recorded during the SVP at Weeks -4, -3, -2, -1 and 0. The mean change of the time adjusted average of hemoglobin from reference value obtained during the SVP (Week -4 up to Week 0) and the value during EEP (Week 17 up to Week 24) was assessed.
Time Frame: Week 17 up to Week 24
Population: ITT population; data missing at the end of the EEP was handled using the last value carried forward method.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
g/dL | -0.3 (1.04)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentration Within the Target Range During EEP
Description: Percentage of participants maintaining hemoglobin concentration within the target range of 10.5 to 12.5 g/dL during EEP (Week 17 to Week 24) was reported.
Time Frame: Week 17 up to Week 24
Population: ITT Population; data missing at the end of the EEP was handled using the last value carried forward method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
percentage of participants | 58.6 [38.9 to 76.5]

4. Secondary Outcome: Mean Time Spent by Participants With Hemoglobin Concentration in the Target Range During the EEP
Description: Mean time spent by participants with hemoglobin concentration within the target range of 10.5 to 12.5 g/dL during the EEP (Week 17 to Week 24) was reported.
Time Frame: Week 17 up to Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
days | 31 (17.2)

5. Secondary Outcome: Percentage of Participants Requiring Any Dose Adjustment
Description: Percentage of participants requiring any adjustment in the dose of study drug during the dose titration period (DTP: Week 1 to Week 16) and EEP (Week 17 to Week 24) was reported.
Time Frame: Week 1 up to Week 16 and Week 17 up to Week 24
Population: ITT Population. Here, 'n' signifies the number of participants evaluable for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
percentage of participants
  DTP (n = 29) | 62
  EEP (n = 26) | 31

6. Secondary Outcome: Percentage of Participants With Red Blood Cell Transfusion During the Study
Description: Percentage of participant who required red blood cell transfusion during the study was reported.
Time Frame: Week 0 up to Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
percentage of participants | 7

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both serious as well as non-serious AEs.
Time Frame: Week 0 up to Week 24
Population: Safety population
Measure: Number; unit: participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 29
participants
  AEs | 22
  SAEs | 9

ADVERSE EVENTS:
Time Frame: Week 0 up to Week 24
Description: Only adverse events with an onset date after the start of medication were included.
Arm/Group | C.E.R.A.
Serious Adverse Events (participants affected / at risk) | 9/29
Other Adverse Events (participants affected / at risk) | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=29)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Diabetic foot infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Renal impairment (Renal and urinary disorders) | 1
Dialysis device insertion (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=29)
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The study was terminated early due to the slow recruitment rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.